CLINICAL TRIAL: NCT02033902
Title: A Global, Postmarketing Observational Safety Study to Evaluate the Safety and Tolerability of Fycompa (Perampanel) as Add-on Therapy in Epilepsy Patients Aged Greater Than or Equal to 12 Years
Status: Completed | Type: Observational
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: E2007-G000-402
Record Dates: First submitted 2013-12-17; First posted 2014-01-13 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2015-11

CONDITIONS: Epilepsy
Keywords: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — perampanel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Perampanel: Perampanel tablets are administered orally according to prescribing information and the treating physician's clinical judgment
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — Perampanel tablets are administered orally according to prescribing information and the treating physician's clinical judgment

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of Fycompa (Perampanel) as an add-on therapy in epilepsy patients aged greater than or equal to 12 years.

DETAILED DESCRIPTION:
This is a global, observational, cohort study in patients with epilepsy. Multiple treating physicians will prescribe perampanel to approximately 500 patients, who then will be observed for approximately 52 weeks.

ELIGIBILITY:
Inclusion Criteria

1. Male or female patients age greater than or equal to 12 years (or as regionally appropriate) at the time of informed consent
2. Patients prescribed perampanel for the adjunctive treatment of epilepsy within 7 days of the Screening Visit
3. Patients who provide informed consent

Exclusion Criteria

1. Participation in another study involving administration of an investigational drug or device whilst participating in this observational study
2. Prior participation in a perampanel clinical study
3. Hypersensitivity to perampanel

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Epilepsy patients prescribed adjunctive treatment in countries where perampanel has received marketing approval. Multiple treating physicians will prescribe perampanel to patients, who then will be observed for approximately 52 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-06-06; Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Number of Treatment Emergent Adverse Events (TEAEs) of interest | Up to 52 weeks and 2 weeks of follow-up
  Assessment of events of dizziness, blurred vision, somnolence, aggression, balance disorders, ataxia, falls, unintended pregnancy, weight gain, suicidality, drug abuse, misuse, dependence, withdrawal, off-label use, skin photosensitivity, unintended pregnancy while taking levonorgestrel-containing contraceptives, and outcomes associated with any suspected drug-drug interaction.

SECONDARY OUTCOMES:
Incidence of unintended pregnancy | Up to 52 weeks
Incidence of off-label use | Up to 52 weeks
Summary scores for the Hospital Anxiety and Depression Scale (HADS) | Screening, Week 52
Number of TEAEs in the patient subpopulations of interest | Up to 52 weeks and 2 weeks of follow-up
  TEAEs observed in the specified subpopulations of patients could also be made in order to get a better understanding of whether any of these particular potential risk factors (e.g., old age, cardiovascular disease) define groups with greater or lesser risk.
Clinical Global Impression of Change | Week 52
  Assessment of disease severity will utilize the Clinical Global Impression of Change (CGI-C) scale at end of treatment to evaluate change in disease status since initiation of treatment.

CONTACTS AND LOCATIONS:
Locations (42):
- Austria (3):
  - Universitatsklinikum Innsbruck, Innsbruck
  - Kepler Universitätsklinikum, Linz
  - Krankenhaus Wien-Hietzing, Vienna
- Belgium (10):
  - Eisai Site# 2405, Battice
  - Hôpital Erasme, Brussels
  - Eisai Site# 2404, Brussels
  - Eisai Site# 2406, Duffel
  - Uz Leuven, Leuven
  - Eisai Site# 2409, Liège
  - Eisai Site# 2403, Ottignies
  - Eisai Site# 2408, Ruddershove
  - Eisai Site# 2407, Woluwe-Saint-Lambert
  - Eisai Site# 2402, Yvoir
- Czechia (6):
  - Eisai Site# 2601, Beroun
  - Eisai Site# 2600, Brno
  - Eisai Site# 2606, Hradec Králové
  - Eisai Site# 2602, Náchod
  - Cerebrovaskularni Poradna S.R.O., Ostrava
  - Eisai Site# 2603, Prague
- Israel (12):
  - Eisai Site# 2013, Beersheba
  - Rambam Medical Center, Haifa
  - Edith Wolfson Medical Center, Holon
  - Kiryat Hadassah, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Western Galilee Hospital, Nahariya
  - Schneider Children's Medical Center Of Israel, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - Eisai Site# 2003, Tel Aviv
  - Eisai Site# 2012, Tel Aviv
  - Eisai Site# 2008, Tel Litwinsky
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Universitetssjukhuset I Linköping, Linköping
- United Kingdom (9):
  - Eisai Site# 1607, Bristol
  - Ninewells Hospital, Dundee
  - Eisai Site# 1611, Lincoln
  - Eisai Site# 1604, London
  - Eisai Site# 1608, London
  - Eisai Site# 1609, London
  - Great Ormond Street hospital, London
  - Eisai Site# 1612, Newcastle
  - Eisai Site# 1606, Truro

REFERENCES:
- [Derived] Maguire M. Response to "Perampanel and pregnancy: Could experience be a gloomy lantern that does not even illuminate its bearer?". Epilepsy Behav. 2022 Apr;129:108654. doi: 10.1016/j.yebeh.2022.108654. Epub 2022 Mar 16. No abstract available. PMID 35305920
- [Derived] Maguire M, Ben-Menachem E, Patten A, Malhotra M, Ngo LY. A post-approval observational study to evaluate the safety and tolerability of perampanel as an add-on therapy in adolescent, adult, and elderly patients with epilepsy. Epilepsy Behav. 2022 Jan;126:108483. doi: 10.1016/j.yebeh.2021.108483. Epub 2021 Dec 23. PMID 34953337